CLINICAL TRIAL: NCT00421460
Title: Phase IV Study of The Therapy of Long-acting Testosterone Undecanoate,1000mg in 4 ml Oily Solution for i.m.Injection(Nebido) as Mono or in Combination With PDE-5 Inhibitors in Hypogonadal Patients With Erectile Dysfunction
Brief Title: The Therapy of Nebido as Mono or in Combination With PDE-5 Inhibitors in Hypogonadal Patients With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Ramathibodi Hospital (Other); Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH 023101
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Hypogonadism; Erectile Dysfunction
Keywords: Nebido in hypogonadism with erectile dysfunction
MeSH Terms: conditions — Hypogonadism; Erectile Dysfunction | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Testosterone Undecanoate,1000mg — duration for 4 injections
  Other Names: Nebido 1000 mg

SUMMARY:
The purpose of this study is to evaluate the response of a treatment with testosterone undecanoate and determine the levels of total and free testosterone in hypogonadal patients with erectile dysfunction.

DETAILED DESCRIPTION:
Hypogonadism is a pathophysiologic and clinical factor in a substantial number of patients with ED,and data indicate that a threshold level of testosterone is necessary for normal erectile function.Testosterone therapy is clearly indicated in hypogonadal patients and is beneficial in other patients with ED and hypogonadism.However,testosterone efficacy as monotherapy for ED could be limited,and combination therapy with testosterone and other ED treatments,such as PDE-5 inhibitors may be valuable in certain subpopulations of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ED over 3 months (specify using IIEF score)
2. Age >= 18 years.
3. Stable sexual relationship
4. With low or low normal serum testosterone level (either total or bioavailable testosterone) TT <= 4 ng/ml and/or BT <= 1 ng/ml
5. Aging Male Symptom scale with total score starting at 37 points (must not replace TT < 4 ng/ml)
6. Eligible subjects who previously took the oral androgen or PDE5 inhibitor must have discontinued their use for 1 month

Exclusion Criteria:

1. Contraindication to treatment with Testosterone according to the SPC
2. Hypersensitivity to the active substances or any of the excipients of Nebido
3. Diagnosed or suspected carcinoma of the prostate or the male breast cancer
4. Past or present liver tumors
5. Acute or chronic hepatic diseases
6. Severe cardiac, hepatic or renal insufficiency
7. History of penile implant or significant penile deformity
8. Diagnosed sleep apnea
9. Polycythemia (Hematocrit >50%)
10. Prolactin >25 ng/ml
11. Organic hypothalamic-pituitary pathology
12. Any unstable medical, psychiatric or drug/alcohol abuse disorder
13. Prostate specific antigen (PSA)>= 4 ng/ml
14. Severe symptomatic benign prostatic hyperplasia (IPSS) sum score >=20)
15. Diabetes mellitus which is uncontrolled (HbAlc level >10%)
16. Epilepsy not adequately controlled by treatment
17. Patients requiring fertility treatment
18. Hypertension which is not adequately controlled on therapy
19. Clinically significant chronic hematological disease which may lead to priapism such as sickle cell anemia, multiple myeloma or leukemia
20. Hypersensitivity to PDE-5 inhibitors
21. Concomitant Medication:

    * Nitrites or Nitric oxide donors
    * Anti-androgens
    * anti-coagulants, with the exception of anti-platelet agents
    * Any of potent inhibitors of cytochrome P-450 3A4:such as HIV protease inhibitors (Ritonavir or Indinavir); Anti-mycotic agent (Itraconazole and Ketoconazole)-topical application allowed; or Erythromycin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Response of treatment for 4 injections at 1 year; score on an IIEF-5 | 4 injections at 1 year for each subject, at 12,30,46 weeks.

SECONDARY OUTCOMES:
Testosterone level | at 6,12,18,36,46 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Apichat Kongkanand, Professor, Principal Investigator — King Chulalongkorn Memmorial Hospital
Locations (3):
- Thailand (3):
  - Siriraj Hospital, Bangkoknoi, Bangkok
  - Ramathibodi Hospital, Rajthevee, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok